CLINICAL TRIAL: NCT02663778
Title: Task Specific Timing and Coordination Exercise to Improve Mobility in Older Adults
Brief Title: Task Specific Timing and Coordination Exercise to Improve Mobility in Older Adults: Program to Improve Mobility in Aging
Acronym: PRIMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jennifer S. Brach, PhD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO14080080
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Gait, Unsteady
MeSH Terms: conditions — Gait Disorders, Neurologic | interventions — Resistance Training; Endurance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard (Active Comparator): The standard arm consists of strength, endurance and flexibility exercises 2 times per week for 12 weeks. Will also receive a physical activity behavioral intervention.
  Interventions: Behavioral: Strength training; Behavioral: Endurance training; Behavioral: Flexibility training; Behavioral: Physical activity behavioral intervention
- Standard-plus (Experimental): The standard-plus arm consists of strength, endurance and flexibility exercises plus task specific timing and coordination exercises to improve gait 2 times per week for 12 weeks. Will also receive a physical activity behavioral intervention.
  Interventions: Behavioral: Strength training; Behavioral: Endurance training; Behavioral: Flexibility training; Behavioral: Task Specific timing and coordination training; Behavioral: Physical activity behavioral intervention

INTERVENTIONS:
Behavioral: Strength training — weight lifting to increase muscle strength
Behavioral: Endurance training — treadmill walking to increase endurance
Behavioral: Flexibility training — stretches to improve flexibility
Behavioral: Task Specific timing and coordination training — stepping and walking patterns to improve timing and coordination of gait
  Arms: Standard-plus
Behavioral: Physical activity behavioral intervention — Intervention to encourage participants to be more physically active

SUMMARY:
This randomized clinical trial targets 248 community-dwelling older adults with impaired mobility (i.e. walking slowly; gait speed < 1.20 m/s). The trial compares a 12 week "standard-plus" program of strength, endurance, flexibility plus task specific timing and coordination training to a standard 12 week strength, endurance and flexibility program. The primary outcome is gait speed at 12 weeks. Secondary and tertiary outcomes represent components of the intervention and measures of activity and participation. Delayed and sustained effects of the intervention are examined at 24 and 36 weeks.

DETAILED DESCRIPTION:
Walking difficulty is common and costly in older adults. While traditional exercise has been shown to promote physical and mental health and may prevent walking difficulty, such exercise has focused on strength and endurance, and has overlooked a critical component of walking ability; the timing and coordination of movement. Aging and disease alter timing and coordination as reflected by slowed neuromotor performance, increased gait variability and reduced smoothness of movement. Task specific timing and coordination exercise that includes practice of smooth coordinated aspects of gait over multiple walking conditions has the potential to improve walking ability greater than a standard program. Our preliminary data suggest that interventions on timing and coordination of gait impact mobility greater than the standard strength and endurance program. The next key step and the objective of this proposal is to combine the two interventions to determine if potential gains in mobility, activity and participation obtained from a standard plus timing and coordination program, are larger than the gains obtained from the standard program alone. Therefore, the primary aim of the proposed project is to evaluate the impact of adding timing and coordination training to standard strength and endurance training on mobility. Secondary aims include examining 1) additional outcomes representing the components of the intervention and measures of activity and participation, 2) the delayed and sustained effects of the intervention, and 3) the effects of the intervention within various other subgroups of interest. This randomized clinical trial in 248 community-dwelling older adults who walk slowly (i.e. < 1.20 m/s) will compare a standard 12 week strength, endurance and flexibility program to a 12 week "standard-plus" program of strength, endurance, flexibility plus task specific timing and coordination training. The primary outcome is gait speed at 12 weeks. We will also examine secondary and tertiary outcomes representing components of the intervention and measures of activity and participation and the delayed and sustained effects at 24 and 36 weeks. The findings from this efficacy trial will provide evidence for the added value of task specific timing and coordination training for promoting walking ability in older adults and will form the basis for future effectiveness trials. Future work includes translation to nonprofessional exercise leaders with the long-term goal to incorporate neurological training into standard exercise programs for health promotion for older adults.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years of age and older
2. Ambulatory without an assistive device or the assistance of another person
3. Usual 4 meter gait speed > 0.60 m/s and < 1.2 m/s
4. Physician clearance to participate in a moderate intensity exercise program
5. Not meeting physical activity recommendations defined as reporting less than 150 minutes of moderate intensity activity per week in the past month.7

Exclusion Criteria:

1. persistent lower extremity pain that is present on most days of the week
2. back pain that is present on most days of the weeks and interferes with walking and activities of daily living or back pain that increases with walking
3. refuse to walk on a treadmill
4. plans to move out of the area in the next 5 years
5. dyspnea at rest or during activities of daily living or use supplemental oxygen (CHF, COPD)
6. any acute illness or medical condition that is not stable according to the approving physician
7. resting systolic blood pressure ≥ 200 mm Hg or diastolic blood pressure ≥ 100 mm Hg or resting heart rate > 100 or < 40 beats per minute
8. diagnosed dementia or cognitive impairment defined as modified Mini-Mental State (3MS) examination <79
9. hospitalized in the past 6 months for acute illness or surgery, other than minor surgical procedures
10. severe visual impairment
11. fixed or fused lower extremity joints such as hip, knee or ankle
12. lower extremity strength <3/5 on manual muscle testing
13. lower extremity amputation
14. progressive movement disorder such as Multiple Sclerosis, Amyotrophic Lateral Sclerosis or Parkinson's disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 353 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Gait speed | 12 weeks
  Usual walking speed over a short distance. A physiologic measure recorded in m/s.

SECONDARY OUTCOMES:
Smoothness of walking | 12, 24, and 36 weeks
  acceleration signal of usual walking. physiologic measure of the acceleration of walking.
gait variability | 12, 24, 36 weeks
  fluctuations in gait characteristics from step to step. physiologic measure of the spatial and temporal gait characteristics
Late Life Function and Disability Instrument - function subscale | 12, 24, and 36 weeks
  Self report measure of function
Late Life Function and Disability Instrument - disability subscale | 12, 24, and 36 weeks
  Self report measure of disability
Lower extremity strength | 12, 24, and 36 weeks
  physiologic measure of leg strength
Lower extremity muscle power | 12, 24, and 36 weeks
  physiologic measure of leg muscle power
Six minute walk test | 12, 24, and 36 weeks
  physiologic measure of walking endurance
Chair sit and reach test | 12, 24, and 36 weeks
  physiologic measure of flexibility
Physical activity | 12, 24, and 36 weeks
  Physiologic measure of physical activity measured using an accelerometer.

OTHER OUTCOMES:
Falls | 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, and 60 weeks
  Self reported falls collected monthly by telephone
Emergency room visits | 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, and 60 weeks
  Self reported emergency room visits collected monthly by telephone
Hospital admission | 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, and 60 weeks
  Self reported hospital admission collected monthly by telephone

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Brach, PhD, PT, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dunlap PM, Crane BM, Perera S, Moored KD, Carlson MC, Brach JS, Klatt BN, Rosso AL. Effects of a Physical Therapist Intervention on GPS Indicators of Community Mobility in Older Adults: A Secondary Analysis of a Randomized Controlled Trial. Phys Ther. 2023 Aug 1;103(8):pzad071. doi: 10.1093/ptj/pzad071. PMID 37364044
- [Derived] Brach JS, Perera S, Shuman V, Gil AB, Kriska A, Nadkarni NK, Rockette-Wagner B, Cham R, VanSwearingen JM. Effect of Timing and Coordination Training on Mobility and Physical Activity Among Community-Dwelling Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2022 May 2;5(5):e2212921. doi: 10.1001/jamanetworkopen.2022.12921. PMID 35604689